CLINICAL TRIAL: NCT03767387
Title: Protocol for Prehabilitation Service Implementation in Catalonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Josep Roca, Clinical Professor, Hospital Clinic of Barcelona
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NEXTCARE-PREHAB
Record Dates: First submitted 2018-12-03; First posted 2018-12-06 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Chronic Disease
Keywords: Prehabilitation; Physical Activity; Integrated Care; Collaborative Self-management
MeSH Terms: conditions — Chronic Disease; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prehabilitation + standard care (Active Comparator): Trimodal Prehabilitation consisting on motivation, personalisation and supervision of physical activity before major surgery
  Interventions: Other: Trimodal Prehabilitation
- Standard care (No Intervention): Standard care before major surgery

INTERVENTIONS:
Other: Trimodal Prehabilitation — Prehabilitation before major surgery consisting of: i) motivational interview to assess patient's adherence profile and to co-design the characteristics of the physical activity program with the patient; ii) personalised program to promote daily physical activity; and iii) supervised high-intensity endurance exercise training program.
  Arms: Prehabilitation + standard care

SUMMARY:
Trimodal prehabilitation consists of a short-term (~ four to six weeks) preventive intervention to: i) enhance aerobic capacity and daily physical activity; ii) nutritional optimization; and, iii) psychological support before a major surgical procedure. The final aim of prehabilitation is to decrease surgical complications and speed-up postoperative functional recovery.

DETAILED DESCRIPTION:
This is a preventive intervention addressed to high risk candidates for major surgical procedures carried out for a period of approximately four weeks before surgery aiming at reducing complications and enhancing post-surgical recovery. It combines: i) high-intensity endurance exercise training and promotion of daily physical activity; ii) nutritional balance; and, iii) psychological support.

The intervention is currently deployed as mainstream service at Hospital Clinic in several types of major surgeries. During fall 2017, three multidisciplinary workshops using a design-thinking approach were carried out to refine the service workflow and to explore the potential for service scalability. The outcomes of the co-design process provided a robust background for the design of a future personalized perioperative care service at regional level covering three phases: prehabilitation, in-patient care, and, post-discharge care.

The current study protocol aims to assess cost-effectiveness of prehabilitation as mainstream service in the ongoing deployment at Hospital Clinic, as well as to generate a roadmap for regional scalability of the service. It is planned as a quasi-experimental case-control study including 500 patients undertaking prehabilitation, as intervention group, and 250 patients following standard conventional care before surgery. The patients will be included from the following type of surgeries (2:1 intervention to control ratio): major digestive surgery (n, 525), lung volume reduction (n, 30), radical cystectomy (n, 30), major cardiovascular surgery (n, 165). Study groups will be made comparable using propensity score matching with the following matching variables: type of surgery, age, sex and adjusted morbidity groups (GMA) scoring.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years old) candidates to colorectal surgery, esophagectomy, gastrectomy, gastric bypass, major liver resection, pancreas resection, lung volume resection, radical cystectomy, cardiac valve surgery or cardiac revascularization.
* Patients at high-risk for surgical complications defined by age > 70 years old and/or American Society of Anesthesiologists 3-4.

Exclusion Criteria:

* Non-elective surgery
* Metastatic disease known preoperatively
* Unstable cardiac or respiratory disease
* Locomotor limitations precluding exercise performance
* Cognitive deterioration impeding adherence to the program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
cost-effectiveness | 4 weeks
  Health care costs

SECONDARY OUTCOMES:
Complications | 4 weeks
  number of complications per patient
Length of stay | 4 weeks
  hospital and intensive care unit length of stay,
Number of hospital readmissions | 4 weeks
  30-day hospital readmissions rate
Number of Emergency room visits | 4 weeks
  30-day emergency room visits rate
Meters achieved in the six-minute walk test | 4 weeks
  Aerobic capacity
Yale Physical Activity Survey (YPAS) | 4 weeks
  Physical activity assessed by the YPAS (Range 0-100) Higher values represent better
Health status assessed by 36-Item Short Form Survey (SF-36) | 4 weeks
  Health status related quality of life (Range 0-100) Higher values represent better
Psychological status assessed by the The Hospital Anxiety And Depression Scale (HAD) | 4 weeks
  Psychological status (Range 0-21) Higher values represent worst

CONTACTS AND LOCATIONS:
Overall Officials: Josep Roca, MD, Principal Investigator — Hospital Clinic
Locations (1):
- Hospital Clinic. Prehabilitation Unit D +34932275747 chernan@clinic.ub.es, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barberan-Garcia A, Ubre M, Roca J, Lacy AM, Burgos F, Risco R, Momblan D, Balust J, Blanco I, Martinez-Palli G. Personalised Prehabilitation in High-risk Patients Undergoing Elective Major Abdominal Surgery: A Randomized Blinded Controlled Trial. Ann Surg. 2018 Jan;267(1):50-56. doi: 10.1097/SLA.0000000000002293. PMID 28489682